CLINICAL TRIAL: NCT06175364
Title: Investigation of the Views of Health Professionals in the Field of Orthotics Prosthetics on Evidence-Based Orthotics Prosthetics Practices
Brief Title: Evidence-Based Orthotics Prosthetics Practices
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Alican AK, Principal Investigator, Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMU-OP-AA-01
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Evidence-Based Practice
MeSH Terms: interventions — Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Professionals in the Field of Orthotics Prosthetics (Other): Health professionals in the field of orthotics and prosthetics generally include orthotic and prosthetic specialists, physiotherapists, rehabilitation specialists, orthopedic surgeons, biomechanics experts, physiologists, and engineers. These professionals specialize in the design, production, application, and rehabilitation of orthoses and prostheses.
  Interventions: Other: Health Professionals in the Field of Orthotics Prosthetics

INTERVENTIONS:
Other: Health Professionals in the Field of Orthotics Prosthetics — Three data collection tools will be used as data collection methods for the research. These data collection tools; demographic information form, Health Sciences Evidence-Based Practice Survey and Information Literacy Self-Efficacy Scale.

SUMMARY:
The main purpose of our research is; The aim of this study is to investigate the views of health professionals in the field of Orthotic Prosthesis in Turkey on Evidence-Based Orthotic Prosthesis Practices. This research is important in revealing the perspective of health professionals in this field on evidence-based orthotic prosthesis applications. No such study has been found in the literature in the field of Orthosis and Prosthesis. In this respect, it aims to bring a new perspective to the literature.

DETAILED DESCRIPTION:
Three data collection tools will be used as data collection methods for the research. These data collection tools; demographic information form, Health Sciences Evidence-Based Practice Survey and Information Literacy Self-Efficacy Scale. Surveys will be sent to participants to be filled out via Google Forms.

Inclusion criteria: Having been working in hospitals, clinics, academic units, etc. in Turkey for at least 6 months. Being able to read and write Turkish. Exclusion criteria; Those who graduated in the field of Orthosis and Prosthesis and work in other clinics and units.

The data will be evaluated in the statistical package program IBM Statistical Package for the Social Sciences Statistics 26.0 (IBM Corp, New York, USA).

To determine the sample size in the study, G*Power 3.1.9.4 software was used to calculate the number of people to take part in the study. The effect size of the study was determined as 134 participants with 80% statistical power and 5% significance level. Our research will be conducted between December 2023 and June 2024.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: Having been working in hospitals, clinics, academic units, etc. in Turkey for at least 6 months.
* Being able to read and write Turkish

Exclusion Criteria:

* Those who graduated in the field of Orthosis and Prosthesis and work in other clinics and units

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Health Sciences Evidence-Based Practice Survey | 2 weeks
  It is a form created to collect participants' information about evidence-based practices in health sciences. The survey is a 10-point Likert scale with a total of 60 items. Main; The scale consists of 3 subheadings: belief-attitude (12 items with total scores ranging from 12 to 120), practice (36 items with total scores ranging from 36 to 360) and barriers-facilitators (12 items with scores ranging from 12 to 120). A higher score indicates a more supportive attitude or behavior towards the implementation of evidence-based practices in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem BOZTAŞ ELVERİŞLİ, Dr.Öğr.Üye., Study Director — MedipolIU
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No